CLINICAL TRIAL: NCT00955994
Title: A Randomized, Double Blind, Parallel Group, Placebo-controlled Study to Evaluate the Effect of On-demand Treatment With Asimadoline in Patients With Irritable Bowel Syndrome Over 4 Weeks
Brief Title: Effect of Asimadoline, a Member of a New Medication Class, on Acute Attacks of Pain in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael Camilleri
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2394-03; IND 67,533
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — asimadoline

INTERVENTIONS:
Drug: asimadoline

SUMMARY:
The treatment of acute pain in patients with irritable bowel symptoms is suboptimal. This is a placebo controlled study of the on demand treatment of pain experienced over a 4 week period in patients with irritable bowel syndrome. Patients will record the severity of pain when they take the study medication and two hours later.

DETAILED DESCRIPTION:
Background:

Asimadoline reduces visceral sensitivity in experimental animal models and has been tested for its effects on gastric sensorimotor function in healthy individuals. It reduces pain sensation in response to distensions that correspond to pressures frequently encountered in the human colon. However, the effects on improvement of pain and gastrointestinal symptoms in individuals with irritable bowel syndrome (IBS) are unclear.

Hypothesis:

The kappa opioid agonist, Asimadoline, reduces pain and discomfort and decreases gastrointestinal symptoms in participants with IBS.

Aim The aim is to compare the effects of Asimadoline (0.5 mg p.r.n, up to 1mg q.i.d.) and placebo on pain and discomfort and other gastrointestinal symptoms in patients with IBS.

Methods:

This is a phase IIB, single center, randomised, double-blind, placebo controlled study of the treatment of pain and discomfort associated with IBS in which study medication or placebo will be administered as required for the relief of these symptoms up to 2 tablets, 4 times per day. After a 2-week run-in period to characterize the nature, frequency and severity of pain to ensure eligibility for the study, participants will treat these pain episodes as the need arises but with strict recommendations on how to self-administer the medication (number, time interval etc?) over a period of 4 weeks. No other pain medications will be permitted during these first 6 weeks (2 weeks run-in, 4 weeks of randomized treatment). During the study, patients will collect daily data which will characterize their pain and other symptoms of IBS, and adequate relief of pain/discomfort. The participants will also keep track of their symptoms and any medications used during a two week observation period after the last dose of medication. A blood sample will be taken and DNA extracted to assess whether IBS patients have single nucleotide polymorphisms in the gene for the kappa receptor.

Anticipated Results and Future Directions:

We anticipate demonstrating that exacerbations of pain in IBS can be effectively reduced by intermittent treatment with the medication, asimadoline. This study will provide preliminary data that will then be used to estimate the sample size required for a phase III program of trials in several centers.

ELIGIBILITY:
Inclusion Criteria

1. Non-pregnant, non-breastfeeding females;
2. 18-65 years old;
3. Established diagnosis of IBS according to Rome II criteria.
4. No alarm indicators on clinical assessment (weight loss of more than 7 kg, bleeding, unexplained recent rectal bleeding uninvestigated by colonoscopy or double contrast barium enema or flexible sigmoidoscopy for the passed 5 years).
5. Females of childbearing potential who are sexually active must be using an acceptable method of contraception for a period of at least one month before the first dose of study medication, continuing through the duration of the study and for one month after the end of the study. Acceptable birth control methods are: surgical sterilization, oral or implanted contraceptive therapy, intrauterine devices and double barrier methods (diaphragm with spermicidal gel or foam or condoms with contraceptive gel or foam). Post-menopausal is defined as >12 months since last menses. Females who are abstinent may participate if they agree to use a double-barrier method of contraception throughout the study should they become sexually active. .
6. Patients must provide written informed consent prior to inclusion in the study.

Exclusion criteria

1. Patients with abdominal pain and discomfort scores less than 40 mm on a VAS or greater scores on less than 4 days out of 14 days during the run-in period (< 30 % of days during the run-in period).
2. Patients with abdominal pain and discomfort scores more than 60 mm on a VAS on more than 10 days out of 14 days during the run-in period (> 70 % of days during the run-in period).
3. Clinically significant abnormal laboratory values at the screening visit
4. Structural or metabolic diseases/conditions that affect the gastrointestinal system. For screening the Bowel Disease Questionnaire 26 which follows in Appendix 1 will be used.
5. Unable to withdraw medications during run-in period that:

   * Alter GI transit including laxatives, antispasmodics, 5-HT 3 antagonists (e.g. alosetron, ondansetron), 5-HT 4 agonists (e.g. tegaserod), triptans (5-HT 1B or 1D agonists), magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, loperamide
   * Analgesic drugs including opiates, NSAID, COX 2 inhibitors
   * Inhibiting CYP 3A4 and 2D6 including carbamazepine, glucocorticoids, phenobarbital, phenytoin, rifampin, systemic antifungal drugs (e.g. ketoconazole)
   * Benzodiazepines NOTE: Low stable doses of antidepressants, thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection and birth control pills or depot injections are permissible.
6. History of positive stool cultures for pathogenic ova or parasites or enteric pathogens within the past 3 months, which has not been successfully eradicated.
7. Female patients who are pregnant or breast-feeding.
8. Clinical evidence (including physical exam, ECG, laboratory tests) and review of the medical history) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study. The Hospital Anxiety and Depression Scale (HADS)33 will be used to exclude patients with significant affective disorders, as well as to determine anxiety and depression scores at the start of the study.
9. Patients known to be hypersensitive to Asimadoline or opioid agonists.
10. Patients who have been previously exposed to Asimadoline.
11. Patients who have participated in another clinical study within the past 30 days.
12. Patients who are considered by the investigator to be alcoholics not in remission or known substance abusers.
13. Previous gastric or intestinal surgery (except appendectomy, cholecystectomy or hysterectomy).
14. Legal incapacity or limited legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Severity of abdominal pain 2 hours after treatment of pain
Average pain reduction within 2 hours after first dose each day ( pain intensity on VAS before and two hours after the first dose on each day with at least moderate pain)
The primary efficacy analysis includes all days with complete data sets for VAS before and two hours after intake of study medication and a before-treatment pain intensity of at least 30 mm on the VAS
For each of these days the pain reduction of the first dose will be calculated: PID (pain intensity difference) = Pain2h ? Pain0h
The average pain reduction on all these days will be calculated by: first, summing up all PID over the treatment period and second, dividing this result by the number of days with pain

SECONDARY OUTCOMES:
Maximum pain during each day
Frequency of bowel movements (number)
Consistency of bowel movements (Bristol stool scale)
Ease of passage
Adequate relief of IBS pain and

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States